CLINICAL TRIAL: NCT05330208
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR-1816 in Healthy Subjects
Brief Title: Single Ascending Dose and Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR-1816 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor internal strategy change.
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SHR-1816-101
Record Dates: First submitted 2022-03-25; First posted 2022-04-15 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: SHR-1816 injection compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: SHR-1816
- Group B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1816 — SHR-1816
  Arms: Group A
Drug: Placebo — Placebo
  Arms: Group B

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR-1816 after single and multiple injection with different dose regimens in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males and infertility females aged between 18 years and 55 years at screening.
2. Male subjects weight ≥50kg, female subjects weight ≥45kg. Body mass index (BMI) in the range of 19-26kg /m2.
3. HbA1c<6.2% at screening.
4. FPG>3.9mmol/L (70mg/dL) and <6.1mmol/L (110mg/dL) at screening
5. Agree to take effective contraceptive methods.
6. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. The following clinical laboratory tests or examination abnormalities exist during the screening period:

1) Any clinically significant lab tests abnormal with one-time retest. 2) ALT and AST were higher than the upper limit of normal value. 3) Subject who has fatty liver disease diagnosed by ultrasound examination. 4) Subject who has abnormal thyroid function. 5) The 12-lead electrocardiogram (ECG) is abnormal and clinically significant, or shows QTcF>450 ms in male and 470 ms in female.

6) Positive infectious diseases screening tests: HBsAg, HCV-Ab, TP-Ig G, HIV-Ab 2. Having any of the following diseases or history:

1. Subject with a history of hypertension or with abnormal vital signs and clinical significance.
2. Subject with a history of life-threatening diseases within the previous 5 years prior to screening.
3. Subject with severe systemic infectious diseases within 1 month prior to screening.
4. Subject with medical history or family history of medullary thyroid cancer, multiple endocrine adenomatosis type 2, and previous history of pancreatitis.
5. Subject with major medical history of heart, liver, kidney, endocrine, digestive, blood, respiratory and genitourinary system or existing diseases of the above systems.

3. Use of any other medicine or other non-drug operations:

1. Prescription drugs, non-prescription drugs, food supplements, vitamins and Chinese herbal medicines within 2 weeks before administration.
2. Subject who received bariatric surgery or procedures, or use of weight-reducing drugs within 3 months prior to administration, or body weight change of more than ±10% within 3 months prior to administration.
3. Drugs that may affect glucose metabolism were used within 1 month before administration.
4. Subject who undergone other gastrointestinal surgery that could lead to malabsorption, or long-term use of drugs that had a direct impact on gastrointestinal motility prior to screening.

4. Any of the following conditions exists:

1. History of allergy to the study drug or any component of it.
2. Treatment with an investigational drug or device within 3 months (or 5 half-lives, whichever is longer) prior to screening.
3. History of regular alcohol consumption in the past week exceeding an average 15g per day and positive alcohol test.
4. More than 5 cigarettes per day or cigarettes in 48 hours before treatment and positive nicotine test.
5. Long time or in 48 hours before treatment drinking for tea, cola, coffee or any other soft drinking within 48 hours.
6. Strenuous exercise in 48 hours before treatment.
7. Subject with known or suspected history of drug abuse or positive urine drug screening test during screening.
8. Unwillingness to comply with lifestyle requirements during the trial.
9. Donate blood within 1 month before screening, or screening trauma or major surgical operation patients who donated blood ≥400 mL or lost blood ≥400 mL within 3 months before the screening.
10. Mentally incapacitated or language impaired subject cannot fully understand or participate in the test process.
11. The investigator assessed the subject's poor compliance or inability to draw blood due to arm vein conditions, or history of needle and blood sickness.

5. Other conditions or laboratory abnormality that may affect trial evaluations associated with study participation reviewed by the investigators.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Number of adverse Events | Day-2 to Day29/Day50
Incidence of hypoglycemic events | Day1 to Day8/Day29
Incidence of reaction of the injection sites | Day1 to Day8/Day29

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of SHR-1816 - AUC0-t | pre-dose, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336 hours post-dose
  AUC0-t, area under the concentration-time curve from time 0 to the time of last quantifiable concentration;
Pharmacokinetic (PK) profile of SHR-1816 - AUC0-inf | pre-dose, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336 hours post-dose
  AUC0-inf, area under the concentration-time curve from time 0 to infinity;
Pharmacokinetic (PK) profile of SHR-1816 - Cmax | pre-dose, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336 hours post-dose
  Cmax, observed maximum concentration;
Pharmacokinetic (PK) profile of SHR-1816 - Tmax | pre-dose, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336 hours post-dose
  Tmax, time of occurrence of Cmax;
Pharmacokinetic (PK) profile of SHR-1816 - Vz/F | pre-dose, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336 hours post-dose
  Vz/F, apparent volume of distribution;
Pharmacokinetic (PK) profile of SHR-1816 - CL/F | pre-dose, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336 hours post-dose
  CL/F, apparent clearance;
Pharmacokinetic (PK) profile of SHR-1816 - t1/2 | pre-dose, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336 hours post-dose
  t1/2, terminal half-life;
Pharmacokinetic (PK) profile of SHR-1816 - MRTinf | pre-dose, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336 hours post-dose
  MRTinf, mean residence time from time 0 to infinity.
Pharmacodynamic (PD) profile of doses of SHR-1816 - fasting blood glucose | Day-1 to Day15/Day29
Pharmacodynamic (PD) profile of doses of SHR-1816 - insulin | Day-1 to Day15/Day29
Pharmacodynamic (PD) profile of doses of SHR-1816 - C-peptide | Day-1 to Day15/Day29
Pharmacodynamic (PD) profile of doses of SHR-1816 - glucagon | Day-1 to Day15/Day29
Pharmacodynamic (PD) profile of doses of SHR-1816 - total GLP-1 | Day-1 to Day15/Day29
Pharmacodynamic (PD) profile of doses of SHR-1816 - active GLP-1 | Day-1 to Day15/Day29
Pharmacodynamic (PD) profile of doses of SHR-1816 - fructosamine | Day-1 to Day15/Day29
PD profile of multiple doses of SHR-1816 - HbA1c | Day-1, Day29
PD profile of multiple doses of SHR-1816 - 7-points glucose profile | Day-1 to Day15/Day29
PD profile of multiple doses of SHR-1816 - weight | Day-1 to Day15/Day29
Immunogenicity | Day1 to Day29/Day50
  Incidence of SHR-1816 antibody formation.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided